CLINICAL TRIAL: NCT01072513
Title: Semen Analysis Following Definitive Treatment of Prostate Cancer With Proton Radiation Therapy Alone
Brief Title: Semen Analysis After Proton Therapy for Prostate Cancer
Acronym: PR08
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UFPTI-0908-PR08
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Semen Analysis, Prostate Cancer, Proton Radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Semen Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semen analysis (Other): Analysis of semen before and after proton radiation therapy.
  Interventions: Other: Semen analysis

INTERVENTIONS:
Other: Semen analysis — Semen analysis before and after proton radiation therapy.

SUMMARY:
The purpose of this study is to evaluate semen for changes following treatment with proton radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of low to intermediate risk prostate cancer and elected to have proton radiation therapy at University of Florida Proton Therapy Institute (UFPTI).

Exclusion Criteria:

* Current use of Flomax, Hytrin, Cardura, Uroxatral, or Rapaflo.
* History of vasectomy.
* Current use of Lupron, Zoladex, Trelstar, Casodex, Eulexin.
* Current use of Avodart or Proscar.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Post treatment sperm count | 12 months after radiation therapy

SECONDARY OUTCOMES:
Compare changes in sperm motility, sperm morphology and semen PH. | 12 months after radiation therapy
  This is composite measure

CONTACTS AND LOCATIONS:
Overall Officials: Bradford S Hoppe, MD, MPH, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Sanda MG, Dunn RL, Michalski J, Sandler HM, Northouse L, Hembroff L, Lin X, Greenfield TK, Litwin MS, Saigal CS, Mahadevan A, Klein E, Kibel A, Pisters LL, Kuban D, Kaplan I, Wood D, Ciezki J, Shah N, Wei JT. Quality of life and satisfaction with outcome among prostate-cancer survivors. N Engl J Med. 2008 Mar 20;358(12):1250-61. doi: 10.1056/NEJMoa074311. PMID 18354103
- [Background] Jang T, Bekelman J, Liu Y, et al. Visits to urologists and radiation oncologists prior to treatment decision making for clinically localized prostate cancer. Journal of Clinical Oncology 2007;25.
- [Background] Grocela J, Mauceri T, Zietman A. New life after prostate brachytherapy? Considering the fertile female partner of the brachytherapy patient. BJU Int. 2005 Oct;96(6):781-2. doi: 10.1111/j.1464-410X.2005.05764.x. PMID 16153199
- [Background] Mydlo JH, Lebed B. Does brachytherapy of the prostate affect sperm quality and/or fertility in younger men? Scand J Urol Nephrol. 2004;38(3):221-4. doi: 10.1080/00365590410025451. PMID 15204375
- [Background] Steinsvik EA, Fossa SD, Lilleby W, Eilertsen K. Fertility issues in patients with prostate cancer. BJU Int. 2008 Sep;102(7):793-5. doi: 10.1111/j.1464-410X.2008.07739.x. Epub 2008 May 16. PMID 18489529
- [Background] King CR, Lo A, Kapp DS. Testicular dose from prostate cyberknife: a cautionary note. Int J Radiat Oncol Biol Phys. 2009 Feb 1;73(2):636-7; author reply 637. doi: 10.1016/j.ijrobp.2008.09.004. No abstract available. PMID 19147028
- [Background] Boehmer D, Badakhshi H, Kuschke W, Bohsung J, Budach V. Testicular dose in prostate cancer radiotherapy: impact on impairment of fertility and hormonal function. Strahlenther Onkol. 2005 Mar;181(3):179-84. doi: 10.1007/s00066-005-1282-1. PMID 15756522
- [Background] Piroth MD, Hensley F, Wannenmacher M, Zierhut D. [Male gonadal dose in adjuvant 3-d-pelvic irradiation after anterior resection of rectal cancer. Influence to fertility]. Strahlenther Onkol. 2003 Nov;179(11):754-9. doi: 10.1007/s00066-003-1108-y. German. PMID 14605745
- [Background] Centola GM, Keller JW, Henzler M, Rubin P. Effect of low-dose testicular irradiation on sperm count and fertility in patients with testicular seminoma. J Androl. 1994 Nov-Dec;15(6):608-13. PMID 7721664
- [Background] Hahn EW, Feingold SM, Simpson L, Batata M. Recovery from aspermia induced by low-dose radiation in seminoma patients. Cancer. 1982 Jul 15;50(2):337-40. doi: 10.1002/1097-0142(19820715)50:23.0.co;2-6. PMID 7083140